CLINICAL TRIAL: NCT05263986
Title: A Phase 1, Open-label, Single-arm Study to Evaluate the Pharmacokinetics and Safety of MRTX849 in Chinese Patients With Advanced Solid Tumors With KRAS G12C Mutation
Brief Title: The Clinical Trial to Evaluate the Pharmacokinetics and Safety of MRTX849 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2312-005
Record Dates: First submitted 2022-01-13; First posted 2022-03-03 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced or Metastatic Solid Tumor
Keywords: KRAS G12C mutation
MeSH Terms: conditions — Neoplasm Metastasis | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): In the 5-day PK lead-in period, patients will receive a single oral dose of 600 mg MRTX849 on Day 1 and there will be no drug administration in the subsequent 4 days. Following the PK lead-in period, patients will receive MRTX849 600 mg BID (an interval of approximate 12 hours between 2 doses) orally in 3-week cycles until disease progression, unacceptable AEs, patient refusal, or death. Dosing schedules may be adjusted depending on safety results.
  Interventions: Drug: MRTX849

INTERVENTIONS:
Drug: MRTX849 — Approximately 18-24 patients to ensure at least 12 PK evaluable patients.
  Subjects will be administered a single oral dose of 600 mg MRTX849 in PK lead in D1, and will start the dosing regimen of 600 mg BID orally from C1D1.

SUMMARY:
This is a phase 1, open-label, single-arm study in Chinese patients with unresectable, locally advanced or metastatic solid tumor with KRAS G12C mutation, for which treatment with curative intent is not available.

Patients must have a documented KRAS G12C mutation determined by tissue or liquid-based local testing.

The PK profile of MRTX849 in Chinese patients will be evaluated after administration of a single and repeat oral doses of 600 mg BID. In the PK lead-in period, blood samples will be collected pre-dose and up to 96 hours post a single oral dose of 600 mg MRTX849. Following this lead-in period, patients will start the dosing regimen of 600 mg BID orally, and blood samples will be collected pre-dose and up to 12 hours after multiple doses of MRTX849 600 mg BID on Cycle 1 Day 8 (C1D8).

Safety including AEs, ECGs, laboratory parameters and vital signs of each patient will be monitored throughout the conduct of the study.

Disease response and progression will be evaluated in accordance with Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diagnosis of a solid tumor malignancy with KRAS G12C mutation.

  2. Unresectable or metastatic disease.

  3. Available therapy:
  1. no available treatment with curative intent,
  2. no available standard-of-care treatment or patient is ineligible or declines treatment.

     4. Presence of measurable or non-measurable disease per RECIST 1.1.

     5. Age ≥ 18 years.

     6. Life expectancy of at least 3 months.

     7. Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy, or investigational agent) and radiation therapy discontinued at least 2 weeks before first dose date.

     8. Recovery from the adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia).

     9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

     10. Laboratory values within the ranges below during the screening period:

  <!-- -->

  1. Absolute neutrophil count ≥ 1,000/mm3 (≥ 1.0 x 109/L)
  2. Platelet count ≥ 100,000/mm3 (≥ 100 x 109/L)
  3. Hemoglobin ≥ 9 g/dL, in the absence of transfusions for at least 2 weeks
  4. Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤ 3 x ULN)
  5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN (if associated with liver metastases, ≤ 5 x ULN)
  6. Creatinine clearance (CrCl) ≥ 60 mL/min.

     11. Women of childbearing potential (WOCBP) or men whose partner is a WOCBP agree to use contraception while participating in this study, and for a period of 6 months following termination of study treatment.

     12. Completed informed consent process, including signing Ethics Committee (EC)-approved informed consent form.

     13. Willing to comply with clinical trial instructions and requirements.

     Exclusion Criteria:
* 1. Use of the treatment known to cause prolonged corrected QT interval (QTc) or with a known risk of Torsades de Pointes that cannot be switched to alternative treatment within 5 half-lives prior to MRTX849 dosing initiation

  2. Use of any drugs or substances including herbal supplements known or suspected to alter MRTX849 absorption, distribution, metabolism, or excretion:
  1. Inhibitors of CYP3A4, CYP2C8, P-glycoprotein (P-gp), or breast cancer resistance protein (BCRP) within 7 days or 5 half-lives, whichever is longer, prior to MRTX849 dosing initiation.
  2. Inducers of CYP3A4 or CYP2C8 within 14 days or 5 half-lives, whichever is longer, prior to MRTX849 dosing initiation.
  3. Proton-pump inhibitors within 7 days or 5 half-lives, whichever is longer, prior to MRTX849 dosing initiation.

     3. Active brain metastases or carcinomatous meningitis. Patients are eligible if brain metastases are adequately treated and patients are neurologically stable for at least 2 weeks prior to study entry without the use of corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).

     4. History of significant hemoptysis or hemorrhage within 4 weeks prior to MRTX849 dosing initiation.

     5. Any of the following cardiac abnormalities:

  <!-- -->

  1. Unstable angina pectoris or myocardial infarction within 6 months prior to

     MRTX849 dosing initiation.
  2. Symptomatic or uncontrolled atrial fibrillation within 6 months prior to

     MRTX849 dosing initiation.
  3. Congestive heart failure ≥ New York Heart Association (NYHA) Class 3 within 6 months prior to MRTX849 dosing initiation.
  4. Prolonged QTc interval > 480 milliseconds.

     6. History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications.

     7. Known human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or C infection. Note that the following are permitted:

  <!-- -->

  1. Patients treated for hepatitis C (HCV) with no detectable viral load;
  2. Patients treated for HIV with no detectable viral load for at least 1 month prior to study entry while on a stable regimen of agents that are not strong inhibitors of CYP3A4; and
  3. Patients with hepatitis B (HBV) receiving prophylaxis against reactivation of hepatitis B (either [HBsAg-positive with normal ALT and HBV DNA <2,000 IU/mL or <10,000 copies/mL] or [HBsAg-negative and anti-HBc-positive]).

     8. Major surgery within 4 weeks prior to MRTX849 dosing initiation.

     9. History of stroke or transient ischemic attack within 6 months prior to MRTX849 dosing initiation.

     10. Known or suspected presence of another malignancy that could be mistaken for the malignancy under study during disease assessments.

     11. Pregnancy. WOCBP must have a negative serum or urine pregnancy test documented within the screening period prior to MRTX849 dosing initiation.

     12. Breast-feeding or planning to breast feed during the study or within 6 months after study treatment with MRTX849.

     13. Any serious illness, uncontrolled intercurrent illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Main PK parameters: Cmax | Approximately 2 weeks after dose initiation
  Maximum plasma concentration (Cmax) after single dose
Main PK parameters: Tmax | Approximately 2 weeks after dose initiation
  Maximum plasma concentration (Tmax) after single dose
Main PK parameters: AUC0-12 | Approximately 12 hours after dose initiation
  Area under the concentration-time curve from time 0 to 12 hours (AUC0-12) after single dose
Main PK parameters: AUC0-t | Approximately 2 weeks after dose initiation
  Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-t) after single dose
Main PK parameters: AUC0-∞ | Approximately 2 weeks after dose initiation
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) after single dose
Main PK parameters: t1/2 | Approximately 2 weeks after dose initiation
  Terminal half-life (t1/2) after single dose
Main PK parameters: CL/F | Approximately 2 weeks after dose initiation
  Apparent clearance (CL/F) after single dose
Main PK parameters: Vz/F | Approximately 2 weeks after dose initiation
  Apparent volume of distribution associated with the terminal phase (Vz/F) after single dose
Main PK parameters: Cmax, ss | Approximately 2 weeks after dose initiation
  Maximum plasma concentration at steady state (Cmax, ss)
Main PK parameters: Tmax, ss | Approximately 2 weeks after dose initiation
  Time to observed maximum plasma concentration at steady state (Tmax, ss)
Main PK parameters: Cmin, ss | Approximately 2 weeks after dose initiation
  Trough concentration (Cmin, ss)
Main PK parameters: Cavg | Approximately 2 weeks after dose initiation
  Average concentration during a dosing interval (Cavg)
Main PK parameters: AUCss | Approximately 2 weeks after dose initiation
  Area under the concentration-time curve at steady state (AUCss)
Main PK parameters: Rac for Cmax and AUCtau | Approximately 2 weeks after dose initiation
  Accumulation ratio (Rac for Cmax and AUCtau)
Main PK parameters: PTR | Approximately 2 weeks after dose initiation
  Peak-to-trough ratio (PTR)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 12 months after dose initiation
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0
Incidence of Treatment-Emergent Serious Adverse Events | Approximately 12 months after dose initiation
  Incidence of Treatment-Emergent Serious Adverse Events as assessed by CTCAE v5.0
Incidence of Treatment-Related Adverse Events | Approximately 12 months after dose initiation
  Incidence of Treatment-Related Adverse Events as assessed by CTCAE v5.0
Incidence of Treatment-Related Serious Adverse Events | Approximately 12 months after dose initiation
  Incidence of Treatment-Related Serious Adverse Events as assessed by CTCAE v5.0
Incidence of abnormal laboratory value | Approximately 12 months after dose initiation
  Incidence of abnormal laboratory value is defined as the proportion of patients who have abnormal laboratory value not prior to the dose initiation of MRTX849

OTHER OUTCOMES:
Objective response rate (ORR) | Approximately 12 months after dosed
  Objective Response Rate (ORR) as assessed by Investigator per RECIST v1.1 Duration of response (DOR)
Duration of response (DOR) | Approximately 12 months after dosed
  Duration of Response (DOR) is defined as the time from radiographic response to disease progression in patients with a best response of CR or PR, assessed per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The first Hospital of Jilin University, Changchun, Jilin
  - Lin Yi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality